CLINICAL TRIAL: NCT06696963
Title: Impact of Time to Initiation of Postoperative Adjuvant Chemotherapy Following Neoadjuvant Chemotherapy on the Prognosis of Locally Advanced Gastric Cancer: a Multi-center Study
Brief Title: Impact of TTC Following Neoadjuvant Chemotherapy on the Prognosis of LAGC
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., M.D. FACS, Fujian Medical University
Other Study IDs: 2024KY039; 2022QNA026 (Other Grant/Funding Number: Fujian Medical University Union Hospital)
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Neoadjuvant chemotherapy; Adjuvant chemotherapy; Time to chemotherapy; survival
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
he present study retrospectively analyzed the clinicopathological data of 524 patients diagnosed with LAGC who underwent D2 radical gastrectomy after NACT between January 2010 and December 2021 at 2 centers. This study was conducted in accordance with the ethical principles outlined in the World Medical Association's Declaration of Helsinki. Informed consent was obtained from all patients and their legal guardians. All procedures were approved by the institutional review board.

DETAILED DESCRIPTION:
This is a retrospective, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* (1) Locally advanced gastric cancer with preoperative clinical staging of cT2-4NxM0 before neoadjuvant chemotherapy. (2) No history of other malignant tumors. (3) No evidence of distant metastasis or invasion of adjacent organs. (4) Underwent gastrectomy after receiving neoadjuvant chemotherapy.

Exclusion Criteria:

* (1) History of prior gastrectomy. (2) History of acute cardiovascular diseases (such as cerebral or coronary artery injuries) within the past three months. (3) Emergency surgery. (4) Did not undergo postoperative adjuvant chemotherapy. (5) Lack of specific information regarding chemotherapy regimens. (6) Loss to follow-up.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally Advnced Gastric Cancer who underwent D2 radical gastrectomy after NACT between January 2010 and December 2021
Sampling Method: Non-Probability Sample
Enrollment: 524 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
3-year all-caused mortality, 3-year Gastric-Cancer Specific Motality | 3 years or 36 months.
  Survival status at 3 years: survival, death, survival with tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China